CLINICAL TRIAL: NCT04785170
Title: Clinical Study to Evaluate Safety and Efficacy of Amino Acid in Healthy Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vedic Lifesciences Pvt. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NN/200602/BAIBA/SA
Record Dates: First submitted 2021-03-03; First posted 2021-03-05 (Actual); Last update posted 2021-05-14 (Actual); Status verified 2021-05

CONDITIONS: Safety and Efficacy
MeSH Terms: interventions — Amino Acids

STUDY DESIGN:
Intervention Model Description: safety and efficacy of amino acid in single arm group of Healthy Individuals.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- amino acid (Experimental): Dose: 1000 mg/day (500 mg/Capsule) Regimen: One capsule after breakfast & one capsule after dinner to be taken with a glass of water.
  Duration: 14 Days
  Interventions: Drug: Amino Acid

INTERVENTIONS:
Drug: Amino Acid — A novel non-protein amino acid secreted by skeletal muscles which aids the cross-talk between skeletal muscles, liver, and adipose tissue at molecular levels. amino acid is generated by catabolism of the branched-chain amino acid valine. Existing literature states, amino acid induces body fat loss by increasing energy expenditure, stimulating free fatty acid (FFA) oxidation in the liver and skeletal muscle cell, and by enhancing oxygen consumption by adipose tissue and hepatocytes. It was observed that amino acid stimulated differentiation of energy storing white adipose tissue preadipocytes to an energy burning "beige" (brown to white) phenotype.

SUMMARY:
In summary, all evidence points in the direction that amino acid supplementation is justified for augmenting desired fat loss associated with physical exercise as an obesity therapy. Nonetheless, the present clinical data concerning oral use of amino acid is insufficient for justifying its usage in humans as questions could arise with regards to its safety. Therefore, the present study was proposed to establish the safety profile of amino acid for human use by evaluating its use at a dose of 1000 mg per day in healthy individuals. The occurrence of adverse events will be monitored and reported as per the Common Terminology Criteria for Adverse Events version 5.0 (CTCAE v5.0), whereas the cardiac safety will be assessed by changes in electrocardiogram parameters, blood pressure, and heart rate. Furthermore, the effect of amino acid consumption on lipid profile will also be assessed by measuring peripheral levels of leptin, adiponectin, total cholesterol, and triglycerides in healthy individuals.

DETAILED DESCRIPTION:
Insufficient physical activity is a global health problem and as per recent literature, approximately one-third of the world's adult population fails to achieve recommended levels of physical activity. An underappreciated primary cause of most chronic conditions is the lack of sufficient daily physical activity. Overwhelming evidence proves the notion that reductions in daily physical activity is primary causes of chronic diseases/conditions and also that exercise is rehabilitative therapy from the inactivity-caused dysfunctions.

There are several underlying mechanisms responsible for exercise-induced benefits such as, organ-to-organ crosstalk that contributes to metabolic homeostasis and affects the inflammatory response related pathways and fibrotic changes. Some of the best recognized beneficial effects of exercise on muscles are mediated by the transcriptional factor peroxisome proliferator-activated receptor gamma coactivator 1-alpha (PGC-1α). Skeletal muscles are highly vascularized tissue and have secretory abilities. Not only muscles release amino acids for fulfilling increased energy demand and to fuel the liver for undergoing gluconeogenesis, but also proteins to mediate inter-tissue crosstalk. Robust research have identified numerous endogenous factors secreted by myocytes (muscle cells) known as myokines or "exercise factor" upon regular exercise via PGC-1α-dependent mechanism. It has been reported that the levels of these myokines are upregulated during aerobic physical exercise.

Amino acid, a novel non-protein amino acid secreted by skeletal muscles which aids the cross-talk between skeletal muscles, liver, and adipose tissue at molecular levels. amino acid is generated by catabolism of the branched-chain amino acid valine. Existing literature states, amino acid induces body fat loss by increasing energy expenditure, stimulating free fatty acid (FFA) oxidation in the liver and skeletal muscle cell, and by enhancing oxygen consumption by adipose tissue and hepatocytes. It was observed that amino acid stimulated differentiation of energy storing white adipose tissue preadipocytes to an energy burning "beige" (brown to white) phenotype. Uptake of plasma nutrients such as glucose, triglycerides (TG)-rich very low-density lipoproteins (VLDL), and FFA by cold-activated brown adipose tissue might be responsible for modulatory effect of amino acid on lipid and glucose metabolism. It is believed that amino acid also exerts its metabolic effects by modulating other circulating signaling molecules such as leptin. amino acid affects lipid metabolism and insulin sensitivity via restoring leptin levels in individuals with leptin deficiency. As about 5-10% of the obese population are low leptin secretor, amino acid might be an ideal intervention for fat loss in such population. It has also been demonstrated that amino acid supplementation activates several "thermogenic programs" similar to those activated by physical exercise. Furthermore, amino acid has been also shown to protect the osteocytes from ROS-induced apoptosis through the MRGPRD and by also maintaining mitochondria integrity. This protective capacity decreases with age as to the down regulation of Mrgprd expression in osteocytes.

ELIGIBILITY:
Inclusion Criteria:

1. Males aged ≥ 18 and ≤ 50 years.
2. Participants with a BMI within the range of ≥ 18.5 kg/m2 to ≤ 29.9 kg/m2
3. Participants deemed healthy by the investigator.
4. Participants willing to abstain from taking any medications that would interfere with outcomes of the study, i.e. lipid lowering medications, gastrointestinal medications, antibiotics, anti-inflammatory drugs, dietary supplements including fiber supplements, prebiotics and probiotics, etc.
5. Able to comply and perform the procedures requested by the protocol (including dietary restrictions, consumption of study treatments, blood sample collection procedures and study visit schedule)
6. Participants who are literate enough to understand the essence of study, are informed about the purpose of the study, and understand their rights.
7. Participants who are able to give written informed consent.

Exclusion Criteria:

1. Presence of type II diabetes mellitus (Indicated by FBS ≥126 mg/dL, with or without drugs)
2. Presence of hypertension (Defined as SBP ≥ 140 mm Hg and/or DBP ≥ 90 mm Hg, with or without drugs)
3. Participants with deranged CMP of severity ≥ grade II as per CTCAE v5.0.
4. Participants with deranged CBC of severity ≥ grade II as per CTCAE v5.0.
5. Participants with ESR < 2 mm/hr or > 15 mm/hr.
6. Participants with heavy alcohol consumption, defined as:

   - For men: More than 14 standard alcoholic drink (SAD)/week or more than 4 SAD in a day.

   (NOTE - A standard alcoholic drink contains approximately 14 grams of alcohol, which is equivalent to 12 ounces of beer (~5% alcohol), 8.5 ounces of malt liquor (~9% alcohol), 5 ounces of wine (~12% alcohol), 3.5 ounces of fortified wine (e.g., sherry or port), or 1.5 ounces of liquor (distilled spirits; ~40% alcohol).
7. Binge drinkers, defined as 5 or more SAD for men, in a 2-hour time frame.
8. Individuals having a history (in past 2 years) of smoking or currently smoking or using any form of smokeless tobacco.
9. Consumption of nicotine, alcohol, coffee, and vigorous physical activity within 48 hours prior to all pre-determined assessment visits.
10. Abnormal Thyroid Stimulating Hormone (TSH) value which is < 0.35 or > 4.94 µIU/mL.
11. Evidence of any infection or inflammatory condition at screening.
12. Participants who have clinically active state of systemic illness which includes but is not limited to cardiovascular, endocrine, immune, respiratory, hepatobiliary, kidney and genitourinary, neuropsychiatric, and gastrointestinal system.
13. Participants diagnosed with any malignancy.
14. Participants having tumors that are being treated or planned for surgery.
15. Participants taking medicines (Prescription, OTC, etc), health functional foods or herbal medicines related to weight reduction within 1 month prior to screening.
16. Participant with significant medication use (inhaled beta agonists, central alpha agonists, hormonal contraceptives, corticosteroid use within three months prior to screening).
17. Participants who participated in another human trial within last 30 days prior to screening.
18. Any condition that could, in the opinion of the investigator, preclude the participant's ability to successfully and safely complete the study or that may confound study outcomes.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2021-02-02 (Actual); Primary Completion 2021-03-26 (Actual); Study Completion 2021-03-26 (Actual)

PRIMARY OUTCOMES:
Adverse Event | 14 Days
  Any Adverse Event / Serious Adverse Event during Treatment Period

CONTACTS AND LOCATIONS:
Locations (1):
- Vedic Life Sciences Pvt. Ltd., Thane, Maharashtra, India

IPD SHARING:
Plan to Share IPD: No